CLINICAL TRIAL: NCT05354284
Title: Physical and Mental Health Among Sexual and Gender Minorities During
Brief Title: Physical and Mental Health Among Sexual and Gender Minorities During Pregnancy, Birth and Postpartum
Status: Active, not recruiting | Type: Observational
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Anna Malmquist, Associated professor, Linkoeping University
Other Study IDs: Reg.nr 2017-499-31
Record Dates: First submitted 2022-02-02; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Sexual and Gender Minorities; Pregnancy Complications; Obstetric Complication; Psychological Trauma
Keywords: Obstetrical complications; Traumatic birth; Mental and physical health; Pregnancy; Birth; Postpartum
MeSH Terms: conditions — Coitus; Pregnancy Complications; Psychological Trauma; Birth Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sexual gender minority people: People self defining Lesbian, Bi-sexual, Transgender, Quer or other are recruited and asked to fill in a questionnaire during pregnancy, three months postpartum and one year later.
  Interventions: Other: online questionnaire

INTERVENTIONS:
Other: online questionnaire — Questionnaire at three timepoints

SUMMARY:
Mental illness increases the risk of adverse birth outcomes (e.g. preterm birth), obstetric complications (e.g. emergency caesarean, birth injuries), and birth trauma. Sexual and gender minority (SGM) people on average experience increased mental illness. Therefore these risks are increased, with risk of prolonged ill health. Despite this, research in this area is scanty. The present project will provide important knowledge for improving the reproductive health of SGM people.

The overall purpose of the project is to increase knowledge about physical and mental health (including fear of childbirth) during pregnancy and postpartum in SGM people. The project has the following aims:

PART I 2017 - 2021Pilotstudy

1. To study fear of childbirth (FOC) among SGM people in Sweden; prevalence and factors associated to FOC
2. To investigate reasons to and consequences of FOC in SGM people

   PART II 2022-2027 Main study
3. To explore whether SGM people in Sweden have an increased incidence of mental illness during and after pregnancy, adverse birth outcomes, obstetric complications and birth trauma.
4. To explore how pre- and postnatal mental health, minority stress, and fear of childbirth correlate to birth outcomes, birth experience, and obstetric complications in SGM people. This is important for identifying specific risk factors for difficult births, and to explore postpartum health effects.
5. To explore in-depth how SGM people have experienced adverse birth outcomes, obstetric complications, and birth trauma, with a specific focus on minority stress and experiences of care during and after pregnancy and childbirth.

DETAILED DESCRIPTION:
Mental illness (fear of childbirth included) during pregnancy increases the risk of adverse birth outcomes (e.g. preterm birth, low birth weight), obstetric complications (e.g. emergency caesarean, instrumental birth, major haemorrhage, perineal laceration), postpartum depression, and postpartum PTSD. Further, social vulnerability, such as belonging to an ethnic minority group, has also been shown to increase the risk of these birth-related complications.

It is also well known that sexual and gender minority (SGM) people (e.g. lesbian and bisexual women, transgender and genderqueer people) on average experience increased mental illness. This is thought to be the consequences of exposure to minority stress.

When stressors related to pregnancy and birth are added to the prolonged minority stress, mental illness increases as a consequence. Previous research shows increased depression, anxiety, and feelings of loneliness and dysphoria during pregnancy, as well as increased risk of postpartum depression, in SGM people.

This indicates that SGM people are at increased risk of adverse birth outcomes, obstetric complications, and traumatic birth experiences, followed by an increased risk of long-term negative effects on their mental and reproductive health. There is very little research on these issues. An American study found that incidence of preterm birth, low birth weight, stillbirth, and caesarean are increased among sexual minority women. However, there are no studies on birth outcomes in gender minority people. Nor are there any publications on obstetric complications or birth trauma in gender or sexual minority people. The present project fills these research gaps.

The data of a pilot study in pregnant SGM people shows an increased prevalence in this group. Fear of childbirth increases the risk of obstetric complications, and is a common reason for requested caesarean. There is unpublished clinical data on caesarean in SGM people that shows a huge overrepresentation in this group. Thus, the study preliminary data indicates that SGM people are at risk of adverse birth outcomes, obstetric complications, and birth trauma, and highlights the need for researching these issues thoroughly.

The overall purpose of the project is to increase knowledge about physical and mental health during pregnancy and postpartum in SGM people, as this knowledge is fundamental for improving the reproductive health of this group. The project has the following aims:

PART I 2017 - 2021Pilot study - data collection completed

1. To study fear of childbirth (FOC) among SGM people in Sweden; prevalence and factors associated to FOC
2. To investigate reasons to and consequences of FOC in SGM people

   PART II 2022-2027 Main study
3. To explore whether SGM people in Sweden have an increased incidence of mental illness during and after pregnancy, adverse birth outcomes, obstetric complications and birth trauma. A register study.
4. To explore how pre- and postnatal mental health, minority stress, and fear of childbirth correlate to birth outcomes, birth experience, and obstetric complications in SGM people. This is important for identifying specific risk factors for difficult births, and to explore postpartum health effects. A longitudinal online survey.
5. To explore in-depth how SGM people have experienced adverse birth outcomes, obstetric complications, and birth trauma, with a specific focus on minority stress and experiences of care during and after pregnancy and childbirth. A qualitative study

The project will be conducted over three years as a collaboration between researchers at two departments at Linköping University: the Department of Biomedicine and Clinical sciences and the Department of Behavioural Sciences and Learning.

Study 1 is a retrospective register study, where data will be analysed during the first two years. Study 2 is a survey study with two measurements within approximately 6 months. It is important that the survey is launched shortly after the onset of the project, to ensure that a sufficient number of participants are included during the project time. Data from Study 2 will be analysed in the last two years of the project. Interviews for Study 3 will be conducted during the first project year and analysed in the second and third year.

This project will generate a knowledge contribution important for the improvement of reproductive health and rights of SGM people giving birth. The present lack of sufficient knowledge in this area is a barrier for healthcare in developing improved and competent care, and in reducing disparities for pregnant and birth-giving SGM people.

The findings of this project will be useful for healthcare professionals within the fields of reproductive and mental health, and will guide the development of accurate and adequate medical and nursing interventions directed at SGM people. Such interventions can be expected to decrease the incidence of adverse birth outcomes, obstetric complications, and birth trauma, improve care when they do occur, and lower the long-term negative health consequences of such sufferings. The project is important for promoting optimal medical and psychosocial outcomes for pregnant SGM people and their children.

ELIGIBILITY:
Inclusion Criteria:

* Self defined LBTQ persons

Exclusion Criteria:

* age under 18, not able to read Swedish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All
Study Population: Pregnant LBTQ people
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
BIrth experience | 3 moths postpartum
  Childbirth Experience Questionnaire (1-4 high levels more positive rating)
Obstetrical complications | 3 moths postpartum
  Self report questionnaire
Mental illness | 3 moths postpartum
  Qualitative interviews
Obstetrical complications | 3 months postpartum
  Qualitative interviews
Fear of child birth | At inclusion
  Wijma Delivery expectancy / experience questionnaire (min 0-max 165. the higher the more severe fear of childbirth)

SECONDARY OUTCOMES:
Depression | At inclusion, 3 months after birth and 1 year after birth
  Hospital anxiety and depression Scale ( 0- 21 points per sub scale, high levels worse condition)
Anxiety | At inclusion, 3 moths after birth and 1 year after birth
  Hospital Anxiety and Depression Scale (0-21/ sub scale, higher levels worse condition.
Traumatic Birth | 3 moths after birth
  City Birth Trauma Scale (0-60 p, high levels means worse condition)
Life quality | At inclusion and 1 year after birth
  Short Form Health Survey 36, SF 36 ( 0-100 high levels better quality of life/ sub scale)
Posttraumatic stress | At inclusion, 3 moths after birth and 1 year after birth
  Impact of event scale 6 items (0-24, high levels more severe condition)

CONTACTS AND LOCATIONS:
Locations (1):
- Linköping University, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No